CLINICAL TRIAL: NCT01373502
Title: International Randomized Comparison Between DES Limus Carbostent and Taxus Drug Eluting Stents in the Treatment of De-novo Coronary Lesions. The NEXT Study.
Brief Title: International Randomized Comparison Between DES Limus Carbostent and Taxus DES in the Treatment of De-novo Coronary Lesions
Acronym: NEXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CID - Carbostent & Implantable Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C20902
Record Dates: First submitted 2010-09-24; First posted 2011-06-15 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Stable Angina; Unstable Angina; Documented Silent Ischemia
MeSH Terms: conditions — Angina, Stable; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DES Limus Carbostent Coronary Stent (Experimental)
  Interventions: Device: DES Limus Carbostent
- Taxus Liberté Coronary Stent (Active Comparator)
  Interventions: Device: Taxus Liberté Stent

INTERVENTIONS:
Device: DES Limus Carbostent — DES Limus Carbostent Carbofilm Coated Coronary Stent
  Arms: DES Limus Carbostent Coronary Stent
Device: Taxus Liberté Stent — Taxus Liberté Coronary Stent
  Arms: Taxus Liberté Coronary Stent

SUMMARY:
The purpose of this study is to demonstrate non-inferiority in terms of safety and efficacy of DES Limus Carbostent compared to the Taxus Liberté in treating de-novo atherosclerotic lesions in native coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient is eligible for percutaneous coronary intervention (PCI) and for surgical revascularization (CABG)
* Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee of the respective clinical site
* Patients with clinical evidence of ischemic heart disease and/or a positive functional study(e.g. stress test); documented stable (CCS I-IV) or unstable angina pectoris (Braunwald class I-II B and C) or documented silent ischemia
* LVEF>30%
* Requires treatment of a single de novo lesion in a native coronary artery in one or two different major epicardial vessels (LAD, LCX or RCA). The second lesion must fit with inclusion/exclusion criteria and must be treated with the same study stent as the first lesion
* Target lesion should be located in a target vessel with a diameter ranging from 3.0 to 3.75 mm
* Target lesion diameter stenosis > 50% and < 100% by visual estimate, with a TIMI flow of ≥ 1
* The target lesion must be appropriately covered (margin of 2.5 mm on both sides of the stent) by one study stent (DES Limus Carbostent or Taxus Liberté, according to the randomization arm). Any occurred dissection of the target vessel must be treated with an additional stent (DES Limus Carbostent or Taxus Liberté, according to the randomization arm)
* Patient that underwent BMS implantation more than 6 months before the enrolment or DES implantation more than 1 year before the enrolment in an other vessel.

Exclusion Criteria:

* Female with childbearing potential or lactating
* Known sensitivity to sirolimus, paclitaxel, the polymeric matrix, stainless steel or cobalt chromium
* Acute Q-wave or non Q-wave myocardial infarction within 72 hours, or presents with CK elevation greater than 2 times upper limit normal associated with elevated CK-MB
* Cardiogenic shock
* Cerebrovascular accident within the past 6 months
* Acute or chronic renal dysfunction (defined as creatinine greater than 2.0 mg/dl)
* Contraindication to aspirin or clopidogrel
* Thrombocytopenia (platelet count less than 100,000/mm³)
* Active gastrointestinal bleeding within the past 3 months
* Known bleeding or hypercoagulable disorder
* Prior anaphylactic reaction to contrast agents or contrast sensitivity that cannot be controlled with pre-medication
* Currently under immunosuppressant therapy
* Currently, or has been treated with either Rapamune or paclitaxel within 12 months of the procedure
* Active infection
* Co-morbidities that could interfere with completion of study procedures, or life expectancy less than 1 year;
* Participating in another investigational drug or device trial that has not completed the primary endpoint or would interfere with the endpoints of this study
* Patient underwent coronary revascularization to any vessel within 30 days
* Patient underwent target vessel revascularization within 6 months
* Target vessel has had prior stent placement
* Presence of two lesions located in the same vascular territory (same major epicardial vessel)
* Prior coronary brachytherapy
* There is a planned target lesion treatment with any technique other than the pre-dilatation balloon angioplasty
* Treatment of more than two lesions is required at the time of enrolment, or is planned within 30 days following enrolment
* Any planned surgery within 6 months after index procedure
* Left main disease greater than 50% diameter stenosis
* Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run off
* Heavily calcified vessel and/or lesion which cannot be successfully predilated
* Target lesion is located or supplied by an arterial or venous bypass graft
* Ostial target lesion or lesion located within 2 mm of a bifurcation
* Target lesion involves a side branch >2.0 mm in diameter with an ostial disease
* Target lesion has TIMI 0 flow
* Target vessel with angiographically visible thrombus or unsuitable for proper stent delivery and deployment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
angiographic efficacy measurement (mm) | 180 days
  in-stent Late Lumen Loss (LLL) measurement by angiography

SECONDARY OUTCOMES:
QCA measurements in-stent and in-segment | 180 days
IVUS measurements | 180 days
Incidence of cardiac death (%) | 30 days, 180 days, 1, 2 , 3, 4 and 5 years
Stent Thrombosis | acute, 30 days, 180 days, 1 year, > 1 year
Acute success (Device and Procedural success) | acute
Incidence of Myocardial Infarction (%) | 30 days, 180 days, 1, 2, 3, 4, 5 years
Incidence of clinically indicated TLR (%) | 30 days, 180 days, 1, 2, 3, 4, 5 years
Incidence of all deaths (%) | 30 days, 180 days, 1, 2, 3, 4, 5 years
Incidence of all repeat revascularization (%) | 30 days, 180 days, 1, 2, 3, 4, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Didier Carrié, Prof, Principal Investigator — Hôpital de Rangueil, Toulouse Cedex 4 - France
Locations (11):
- Belgium (2):
  - Academisch Ziekenhuis Middelheim, Antwerp
  - Ziekenhuis Oost Limburg, Genk
- France (4):
  - Clinique les Franciscaines, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - Clinique Saint-Hilaire, Rouen
  - Hôpital de Rangueil, Toulouse
- Germany (2):
  - Medizinisches Versorgungszentrum, Hamburg
  - Krankenhaus der Barmherzigen Brüder, Trier
- Italy (3):
  - Azienda Ospedaliera Careggi, Florence
  - Istituto di Fisiologia Clinica del CNR, Massa
  - Ospedale S. Camillo, Roma

REFERENCES:
- [Derived] Carrie D, Berland J, Verheye S, Hauptmann KE, Vrolix M, Violini R, Dibie A, Berti S, Maupas E, Antoniucci D, Schofer J. A multicenter randomized trial comparing amphilimus- with paclitaxel-eluting stents in de novo native coronary artery lesions. J Am Coll Cardiol. 2012 Apr 10;59(15):1371-6. doi: 10.1016/j.jacc.2011.12.009. Epub 2012 Jan 25. PMID 22284328